CLINICAL TRIAL: NCT03181815
Title: Efficacy and Safety of Cladribine in Combination With G-CSF, Low-dose Cytarabine and Aclarubicin in Patients With Refractory/Relapsed Acute Myeloid Leukemia: a Phase 2 Clinical Trial
Brief Title: Cladribine in Combination With CAG in Patients With Refractory/Relapsed Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Liang Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-CAG in AML
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Acute Myeloid Leukemia; Relapse Leukemia
Keywords: CLADRIBINE; ACUTE MYELOID LEUKEMIA
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cladribine; Granulocyte Colony-Stimulating Factor; Aclarubicin; aclacinomycins; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): The patients in this arm will receive C-CAG regimen for salvage treatment,detailed as following: Cladribine 5mg/㎡，d1-5；G-CSF 300ug,d0-9; aclarubicin 10mg,d3-6;cytarabine 10mg/㎡ q12h, SC, d3-9;4 weeks a cycle
  Interventions: Drug: Cladribine; Drug: G-CSF; Drug: Aclarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Cladribine — 5mg/㎡ d1-5
  Other Names: cladribine injection
Drug: G-CSF — 300ug d0-9
  Other Names: granulocyte
Drug: Aclarubicin — 10mg d3-6
  Other Names: Aclacinomycin
Drug: Cytarabine — 10mg/㎡ q12h SC d3-9
  Other Names: Ara-C

SUMMARY:
The vast majority of patients with AML will die of the disease, and no standard chemotherapy regimen were defined for patients with relapsed/refractory AML. Previous studies have confirmed the efficacy of cladribine in the treatment of AML, both de novo or relapse/refractory AML. Our previous experience has shown that Cladribine in combination of CAG (G-CSF priming, low dose cytarabine, and aclarubicin) are effective with tolerable toxicity profiling.Thus, this phase 2 clincial trial is going to evaluate the efficacy and safety of cladribine in combination with G-CSF, low-dose cytarabine and aclarubicin (C-CAG) in patients with refractory/relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
AML is most common in the elderly patients, who can not tolerate the intensified treatments. The vast majority of patients with AML will die of the disease, and no standard chemotherapy regimen were defined for patients with relapsed/refractory AML. Previous studies have confirmed the efficacy of cladribine in the treatment of AML, both de novo or relapse/refractory AML. Our previous experience has shown that Cladribine in combination of CAG (G-CSF priming, low dose cytarabine, and aclarubicin) are effective with tolerable toxicity profiling.Thus, this phase 2 clincial trial is going to evaluate the efficacy and safety of cladribine in combination with G-CSF, low-dose cytarabine and aclarubicin (C-CAG) in patients with refractory/relapsed acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Clinical diagnosis of Relapsed/Refractory AML (non-APL);
* ECOG performance status (PS) score 0-3;
* AST and ALT <=2.5 times the institutional ULN;
* Total bilirubin <=2.0 times the institutional ULN
* Serum creatinine<2.0 times the institutional ULN;
* Subjects should take effective contraceptive measures，and serum or urine pregnancy tests must be negative during the screening and study periods in women subjects;
* Patients should understand the disease and voluntarily receive the study regimen and follow-up.

Exclusion Criteria:

* Concurrent diagnosis of tumors other than AML, with exclusion of superficial bladder cancer, basal cell and squamous cell carcinoma, cervical intraepithelial neoplasms (CIN), prostatic intraepithelial neoplasms(PIN);
* Active viral or bacterial infection that would impair the ability of the subject to receive protocol therapy;
* Concurrent autoimmune hemolytic anemia or immune thrombocytopenia;
* Subjects suffered from AIDS，active hepatitis B or C virus infection; 垫·Dementia or altered mental status that would prohibit the understanding or rendering of informed consent;
* Be allergic to any component of C-CAG regimen;
* Subjects ever exposed to cladribine or CAG-based regimen.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR) rate | Bone marrow aspiration will be done within 2 weeks after blood cell count recovery (about 4 weeks after initiation of C-CAG treatment)
  Less than 5% of blast cells in bone marrow aspiration is defined as CR.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From initiation of C-CAG treatment to end of the study (about within 3 months since enrollment)
  The hematologic toxicities and non-hematologic toxicities will be graded according to CTCAE version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Liang Wang, M.D., Principal Investigator — Sun Yat-sen Univerisity
Locations (1):
- Liang Wang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided